CLINICAL TRIAL: NCT03326310
Title: Phase I Study of MEK Inhibitor Selumetinib in Combination With Azacitidine in Patients With Higher Risk Chronic Myeloid Neoplasia: MDS, MDS/MPNs, and Myelofibrosis
Brief Title: Selumetinib and Azacitidine in High Risk Chronic Blood Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-0774
Record Dates: First submitted 2017-10-13; First posted 2017-10-31 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Chronic Myeloid Leukemia; Myelofibroses
Keywords: Chronic Myeloid Leukemia; Myelofibrosis; selumetinib; azacitidine
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Primary Myelofibrosis | interventions — Azacitidine; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azacitidine and selumetinib (Experimental): Subjects will receive azacitidine subcutaneously on days 1-7. Selumetinib will be administered on days 8-21. Subjects will continue on this schedule in cycles of 28 days duration in the absence of disease progression.
  Interventions: Drug: Azacitidine; Drug: Selumetinib

INTERVENTIONS:
Drug: Azacitidine — Patients will receive azacitidine 75 mg/m2 as a subcutaneous injection on days 1-7. The dose of azacitidine 75 mg/m2 will remain unchanged, unless a dose reduction is required based on toxicities (dose level -1 = selumetinib 50 mg PO twice daily and azacitidine 50 mg/m2).
  Subjects will continue on this schedule in cycles of 28 days duration in the absence of disease progression
  Other Names: Vidaza
Drug: Selumetinib — Patients will receive selumetinib administered by mouth on days 8-21. The starting dose cohort (dose level 1) will receive selumetinib 50 mg PO twice daily on days 8-21. Subsequent planned doses include selumetinib 75 mg PO twice daily (dose level 2) and selumetinib 100 mg PO twice daily (dose level 3). Subsequent dose levels will only be given once the prior dose level has shown acceptable safety.
  Subjects will continue on this schedule in cycles of 28 days duration in the absence of disease progression.
  Other Names: AZD6244

SUMMARY:
This is a phase I, open-label, dose-escalation study to determine the MTD of selumetinib when combined with the standard dose of azacitidine. Treatment will begin within 28 days of screening procedures. Treatment will continue indefinitely, provided that the patient continues to derive benefit. A patient will be taken off study for reasons described in detail in section 3.12 including disease progression, unacceptable toxicity, inter-current illness, withdrawal of consent, or at the discretion of the investigator. Patients will be followed for 12 weeks after the last dose of study drug, until any study treatment related toxicities have stabilized, or until death. The total duration of the study is expected to be approximately 24 months.

DETAILED DESCRIPTION:
This is a phase I, open-label, dose-escalation study to determine the MTD of selumetinib when combined with the standard dose of azacitidine. For the purposes of DLT assessment, subjects will be stratified into 2 cohorts- cohort A will include subjects with MDS and MDS/MPN; cohort B will include subjects with myelofibrosis. Dose escalation will proceed independently in each of these cohorts. Determination of MTD will thus also proceed independently within each cohort. Three dose levels of selumetinib are planned for evaluation. Dose escalation will follow a 3+3 study design. Patients will be enrolled sequentially and stratified according to disease type as outlined above. An increased dose level will only open to accrual once at least 3 patients have been treated at the lower dose, followed for the defined DLT observation period (28 days, see section 2.8 below), and the lower dose level has been deemed safe.

The 3+3 dose escalation algorithm will proceed as follows:

1. If 0/3 patients develop a DLT at a dose level, escalate to the next dose level.
2. If 1/3 patients develops a DLT at a dose level, enroll 3 additional patients at that dose level.

   1. At that dose level, if 1/6 patients develops a DLT, escalate to the next dose level.
   2. If ≥2/6 patients develop a DLT, that dose level will be determined to be too toxic.
3. If 2-3/3 patients develop a DLT at a dose level, that dose level will be determined to be too toxic.
4. Six patients will be treated at the MTD.

   1. If the study progresses to dose level 3 with 0/3 patients experiencing a DLT, an additional 3 patients will be enrolled at that dose level to gain additional information regarding toxicity.
   2. If a dose level is determined to be too toxic and the next lower dose level only included 3 patients, an additional 3 patients will be treated at the lower dose level to confirm tolerability.
5. If no patients have a DLT reported at dose level 3, that will be defined as the MTD and the dose will not be escalated above that level.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be met:

* Age greater than or equal to 18 years of age
* Histologic confirmation of one of the following:

  a. MDS fulfilling all the criteria below: i. International Prognostic Scoring System (IPSS) intermediate-2 or high risk MDS; or Revised International Prognostic Scoring System (IPSS-R) intermediate, high, or very high risk MDS ii. - relapsed/refractory disease iii. Requiring therapy based on the presence of one or more cytopenias (Hb <10 g/dL and/or red cell transfusion dependence, platelets- <50,000/μL, or ANC <1,000/ μL) or excess blasts (≥5% in the peripheral blood or bone marrow).

  b. MDS/MPN as defined by the WHO criteria, including CMML, atypical CML, and MDS/MPN-Unclassifiable fulfilling the criteria listed below i. relapsed/refractory disease ii. Requiring therapy based on the presence of one or more cytopenias (Hb <10 g/dL and/or red cell transfusion dependence, platelets <50,000/μL, or ANC <1,000/ μL), excess blasts (≥5% in the peripheral blood or bone marrow), or palpable splenomegaly iii. or previously untreated subsets (e.g atypical CML, MDS/MPN unclassifiable) requiring therapy as defined above and in whom no approved therapies exist.

  c. Myelofibrosis, including primary myelofibrosis, post-polycythemia vera myelofibrosis, or post-essential thrombocythemia myelofibrosis fulfilling the criteria listed below: i. Intermediate-2 or high risk disease according to the Dynamic International Prognostic Scoring System (DIPSS) classification ii. refractory or intolerant to JAK inhibitor therapy, or deemed - ineligible for ruxolitinib therapy due to pre- existing cytopenias (thrombocytopenia <50,000/uL, anemia hemoglobin <9g/dL or red cell transfusion dependence).Requiring further therapy based on the presence of one or more cytopenias (Hb <10 g/dL and/or red cell transfusion dependence, platelets <50,000/μL, or ANC <1,000/μL), excess blasts (≥5% in the peripheral blood or bone marrow), or palpable splenomegaly
* No history of prior exposure to a MEK inhibitor
* ECOG performance status of ≤ 2
* Adequate renal function, defined as serum creatinine ≤ 1.5 x ULN or creatinine clearance >30 mL/min based on the Cockroft-Gault equation: (140 - Age) x (weight in kg) x (0.85 if female) / 72 x serum creatinine
* Adequate liver function, defined as conjugated bilirubin ≤ 2 x ULN as well as aspartate transaminase (AST) and alanine aminotransaminase (ALT) ≤ 3 x ULN
* Patients must be at least 2 weeks from major surgery, radiation therapy, participation in other investigational trials and must have recovered from clinically significant toxicities of these prior treatments
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment
* Female and male patients must use an effective contraceptive method during the study and for at least 6 months thereafter
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

Patients are excluded if any one of the following is present:

* Receipt of any anti-cancer therapy within 14 days prior to study entry, with the exception of hydroxyurea. If clinically indicated in order to keep WBC <30,000/uL, hydroxyurea may be continued through the first cycle.
* Concurrent active malignancy, with the exception of early stage basal cell or squamous cell skin cancer
* Active cardiac conditions, including any of the following:

  1. Uncontrolled hypertension (BP >150/95 mmHg despite medical therapy)
  2. Acute coronary syndrome within 6 months prior to starting treatment
  3. Uncontrolled angina despite medical therapy
  4. Symptomatic heart failure (NYHA class II-IV despite medical therapy)
  5. Baseline LV EF <50% measured by either echocardiography or MUGA scan
  6. Severe valvular heart disease
  7. Atrial fibrillation with ventricular rate >100 bpm on EKG at rest.
* Ophthalmologic conditions, including any of the following:

  1. Current or past history of central serous retinopathy
  2. Current or past history of retinal vein occlusion
  3. Intraocular pressure (IOP) >21 mmHg or uncontrolled glaucoma
* Any uncontrolled concurrent illness that, in the judgment of the investigators or treating physician, may put the patient at undo risk including but not limited to active infection, symptomatic cardiac or pulmonary disease, ventricular arrhythmia, or psychiatric illness.
* Pregnant or lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-09-04 (Actual); Primary Completion 2027-09-04 (Estimated); Study Completion 2027-09-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | Up to 24 months.
  To determine the maximum tolerated dose (MTD) of selumetinib when combined with azacitidine and measure any toxicities that may arise.

SECONDARY OUTCOMES:
Time to completion of next generation sequencing panel. | From the start of treatment to the record of patient death from any cause, or 100 months, whichever comes first.
  To assess the feasibility of prospectively screening patients for RAS pathway activating mutations by next generation sequencing at our center in the context of a clinical trial.
Rate of overall response. | From the start of treatment to the first record of response, up to 100 months, whichever comes first.
  Calculated by complete response + partial response + hematologic improvement.
Rate of symptom response. | From the start of treatment to the first record of symptom response, up to 100 months, whichever comes first.
Rate of overall survival. | From the start of treatment to the date of death, not to exceed 100 months, whichever comes first.
Rate of progression free survival. | From the start of treatment to the first record of disease progression or the date of death, not to exceed 100 months, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Olatoyosi Odenike, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States